CLINICAL TRIAL: NCT06610344
Title: Preliminary Investigation of Β-hydroxybutyrate Supplementation for Lymphoma Patients Receiving Anti-CD19 CAR T-cells
Brief Title: BHB & CAR-T for Lymphomas
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UPCC 41424; IRB#856611 (Other: University of Pennsylvania IRB)
Record Dates: First submitted 2024-09-20; First posted 2024-09-24 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-02

CONDITIONS: Large B-cell Lymphoma
MeSH Terms: interventions — beta-hydroxybutyrate-1,3-butanediol monoester; Ketones

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- R-1,3-Butanediol (Experimental): Participants will take 35mL of HVMN Ketone-IQ by mouth three times daily, with each dose containing 10 grams of R-1,3-Butanediol.
  Interventions: Dietary Supplement: R-1,3-Butanediol

INTERVENTIONS:
Dietary Supplement: R-1,3-Butanediol — R-1,3-Butanediol 35 mL
  Other Names: Ketone

SUMMARY:
The aim of this study is to assess the feasibility of β-hydroxybutyrate (BHB) supplementation in individuals who are receiving therapy for lymphoma with standard-of-care anti-CD19 CAR T-cells (CAR-T) to determine whether BHB supplementation is safe and tolerable in this patient population. Additionally, this study will determine whether BHB supplementation leads to changes the gut microbiome and peripheral blood mononuclear cells (PBMCs). BHB supplementation will be performed through oral administration of HVMN Ketone-IQ, a commercially available BHB supplement, with an active ingredient of R- 1,3-Butanediol, which is converted to BHB.

ELIGIBILITY:
Inclusion Criteria:

* Age of 18 years or older
* History of pathologically-confirmed large B-cell lymphoma (LBCL)
* Planned treatment with a commercially available anti-CD19 CAR-T product (Yescarta or Kymriah)
* Eligible for and with adequate organ function (investigator discretion) and performance status (ECOG PS 2 or less) for standard of care, anti-CD19 CAR-T
* Not enrolled on a clinical trial of bridging therapy prior to CAR-T
* Patients must have a PET/CT scan (preferred), diagnostic CT scan, or MRI with at least one bi-dimensionally measurable lesion (≥ 1.5 cm for nodal lesions or ≥ 1cm for extra- nodal lesions in largest dimension by low-dose computerized tomography [CT] scan with FDG-uptake ≥ liver) documented prior to leukapheresis for CAR-T manufacturing
* Resolution of toxicities from prior therapy to a grade that does not contraindicate trial participation in the opinion of the investigator
* Can provide informed consent
* Willing to comply with all study procedures and available for the duration of the study

Exclusion Criteria:

* Subject is pregnant or breast feeding
* History of allergy to energy drinks
* History of inflammatory bowel disease
* History of type 1 diabetes mellitus or requirement for insulin
* History of chronic kidney disease with an eGFR < 30 mL/min/1.73m2
* Additional second primary malignancy for which the subject is receiving active therapy or that will impede the ability of the investigator to assess lymphoma response

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Estimated)
Dates: Start 2025-01-07 (Actual); Primary Completion 2025-10-15 (Estimated); Study Completion 2026-10-15 (Estimated)

PRIMARY OUTCOMES:
Safety and tolerability | From CART infusion to day 28 visit after CART
  Assess number and severity of adverse events as well as number of patients who complete treatment

SECONDARY OUTCOMES:
Changes in gut microbiome | prior to BHB administration to day 28 visit after CART
  compare changes in stool microbiome diversity assessed by stool 16S rRNA gene sequencing, metabolomics, qPCR
Changes in peripheral blood mononuclear cells | prior to BHB administration to day 28 visit after CART
  compare changes in number and phenotype using flow cytometry, single cell RNAseq, qPCR

CONTACTS AND LOCATIONS:
Overall Officials: Elise Chong, MD, Principal Investigator — Abramson Cancer Center at the University of Pennsylvania
Locations (1):
- Abramson Cancer Center at University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Undecided
It is not yet known if there will be a plan to make IPD available. Explanation: currently under discussion regarding logistics of sharing, data to be shared, and how to access. Some IPD, likely CSR, will be shared after publication. We will finalize a plan by 3/2025